CLINICAL TRIAL: NCT03805282
Title: Intravenous Lidocaine Continuous-infusion to Supress of Cough Reflex During Anesthesia Emergence: Dose-finding Adaptive Trial
Brief Title: Intravenous Lidocaine to Supress of Cough Reflex During Anesthesia Emergence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of Anesthesiology, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LidoTosse
Record Dates: First submitted 2017-12-26; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Cough
Keywords: general anesthesia; cough; anesthesia emergence; lidocaine
MeSH Terms: conditions — Cough | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Four parallel groups will be studied:
  * Female > 60 years old
  * Male > 60 years old
  * Female 18 to 60 years old
  * Male 18 to 60 years old
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A study participant who will not participate during assessment of the main outcome will prepare the drug solutions to be infused at 10ml/h accordingly to the response of the previous patient and to the dose calculated for the next patient. The participant who will verify the main outcome during anesthesia emergence will not know the dose the patient is receiving. Participants will not be informed of the dose they will receive. The outcomes assessor will not handle individual data and statistical analysis plan was developed in advance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Female 18 to 60 years old (Experimental): This adaptive dose-finding group will receive continuous infusion lidocaine using the biased coin method for finding the 95% effective dose (ED95%) for cough suppression. All patients will also receive remifentanil 0.025mcg/kg.h during emergence.
  Interventions: Drug: Lidocaine
- Male 18 to 60 years old (Active Comparator): This adaptive dose-finding group will receive continuous infusion lidocaine using the biased coin method for finding the 95% effective dose (ED95%) for cough suppression. All patients will also receive remifentanil 0.025mcg/kg.h during emergence.
  Interventions: Drug: Lidocaine
- Male > 60 years old (Active Comparator): This adaptive dose-finding group will receive continuous infusion lidocaine using the biased coin method for finding the 95% effective dose (ED95%) for cough suppression. All patients will also receive remifentanil 0.025mcg/kg.h during emergence.
  Interventions: Drug: Lidocaine
- Female > 60 years old (Active Comparator): This adaptive dose-finding group will receive continuous infusion lidocaine using the biased coin method for finding the 95% effective dose (ED95%) for cough suppression. All patients will also receive remifentanil 0.025mcg/kg.h during emergence.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Continuous infusion, variable dose of lidocaine.
  Other Names: Xylocaine

SUMMARY:
Introduction: Although inflating tracheal cuff using lidocaine is effective for cough suppression, it may pressure tracheal cuff too much. Intravenous continuous infusion of lidocaine has emerged recently for most general anesthesia in the context of opioid-sparing anesthesia for cancer, but the 95% effective dose (ED95) for cough suppression during anesthesia emergence is not determined yet. Objective: the objectives of this study are to determine the ED95 of continuous infusion lidocaine for suppressing cough reflex during extubation by sex and age group.

DETAILED DESCRIPTION:
Ideal patient weight in kg will be considered.

Initial dose will be 0.5mg/kg.h and dose-change steps of 0.5mg/kg.h will occur depending on the incidence of emergence cough in the previous patient of the same group:

* It will increase if coughed in a probability of 95%
* It will decrease if not coughed in a probability of 5%.
* It will remain the same otherwise. Maximum dose will be 3mg/kg.h. All patients will receive remifentanil 0.025mcg/kg.min continuous infusion until extubation.

Patients groups will be determined by sex and age group (18-60 or >60 years old), therefore, four independent groups will be studied:

* Female 18 to 60 years old
* Male 18 to 60 years old
* Female > 60 years old
* Male > 60 years old

ELIGIBILITY:
Inclusion Criteria:

* Understands study risks and benefits, signs informed consent.
* Not pregnant.
* Not an airway surgery
* No acute or chronic respiratory disease.
* Non smoker
* No chronic cough

Exclusion Criteria:

* Any protocol violation.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cough during anesthesia emergence | Anytime during anesthesia emergence, before extubation.
  Dichotomic variable, true if any cough is detected from anesthesia weaning to extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
we will make IPD available in www.anestesiologiaunb.com.br
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In a year following the study
Access Criteria: Open
URL: http://www.anestesiologiaunb.com.br